CLINICAL TRIAL: NCT04320901
Title: Comparative Analysis Between Harmonic Versus LigaSure in Transoral Endoscopic Thyroidectomy: A Randomized Controlled Trial
Brief Title: Energy Device Study in Transoral Endoscopic Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Jin Wook Yi, Assistant Professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01-033
Record Dates: First submitted 2020-03-20; First posted 2020-03-25 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Thyroid Nodule; Thyroid Cancer
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms | interventions — Second Harmonic Generation Microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Harmonic (Experimental): Endoscopic procedure will be done by Harmonic ACE7+
  Interventions: Device: Harmonic
- Ligasure (Experimental): Endoscopic procedure will be done by Ligasure
  Interventions: Device: Ligasure

INTERVENTIONS:
Device: Ligasure — Ligasure™ Maryland Jaw Laparoscopic Sealer/Divider 37cm
  Arms: Ligasure
Device: Harmonic — Harmonic ACE 7+
  Arms: Harmonic

SUMMARY:
Open label randomized controlled study, for Harmonic versus Ligasure in transoral endoscopic thyroid surgery.

DETAILED DESCRIPTION:
* This is a prospective randomized controlled study. The principal investigator or another clinical investigator in charge will individually inform the patients about the study, on the day before surgery.
* When informed consent is obtained, an investigator in charge of randomization only, will randomize the patients.
* According to randomization, the experimental group will Ligasure and the control group will use Harmonic ACE 7+. Other than the randomized use of energy devices, the protocol for TOETVA is performed as usual.
* Operation time (from insertion of the laparoscopic camera to removal of the camera), number of times the camera was cleaned, intraoperative blood loss will recorded.
* Postoperative hospital stay, visual analog pain scale, blood cell count and inflammatory parameters, postoperative drain amount will recorded.
* Complications of thyroid surgery (vocal cord dysfunction, hypoparathyroidism) are compared for safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who planned to transoral endoscopic thyroidectomy
* Age between 20 to 70
* Voluntarily consenting to the study and study agreement
* No local invasion or distant metastasis
* Normal vocal cord function in laryngoscopic exam
* No significant abnormalities in preoperative laboratory tests

Exclusion Criteria:

* Take aspirin or antiplatelet drugs within 7 days before admission
* Uncontrolled hypertension, diabetes, chronic renal failure, or coagulation disease
* History of cardiovascular disease (angina pectoris, heart failure, myocardial infarction, history of coronary artery disease, stroke, transient ischemic attack)
* Substance abuse and alcohol abuse
* History of esophageal and airway diseases
* Patient was participated in other clinical trials within 30 days
* History of neck irradiation or surgery
* History of severe drug allergies
* Pregnant or lactating women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Operation time | During the procedure
  Surgery time during the thyroid lobectomy
Camera cleaning frequency | During the procedure
  Numbers of camera cleaning during the lobectomy
Blood loss | During the procedure
  Estimated blood loss during the lobectomy

SECONDARY OUTCOMES:
Pain score | Postoperative 1st and 2nd days
  visual analogue scale, ranged from 0-10 (0: no pain, 10: maximal pain)
Drain amount | Postoperative 1st and 2nd days
  24-hour drain amount (ml/day)

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

REFERENCES:
- [Derived] Park SY, Shin MH, Hwang YM, Choi YS, Yi JW. Comparative analysis between ultrasonic shears versus advanced bipolar device in transoral endoscopic thyroidectomy: a randomized controlled trial. Gland Surg. 2023 Sep 25;12(9):1191-1202. doi: 10.21037/gs-23-227. Epub 2023 Sep 18. PMID 37842523